CLINICAL TRIAL: NCT05600816
Title: CHOMP: SurmodiCs Pounce Venous THrOMbectomy System Post Market Clinical Follow Up Study
Brief Title: SurmodiCs Pounce Venous THrOMbectomy System Post Market Clinical Follow Up Study
Acronym: CHOMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUR21-001
Record Dates: First submitted 2022-02-09; First posted 2022-11-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Vascular Occlusive Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pounce Venous Thrombectomy System (Other): Subjects admitted for endovascular thrombus removal using the Pounce Venous Thrombectomy System
  Interventions: Device: Pounce Venous Thrombectomy System

INTERVENTIONS:
Device: Pounce Venous Thrombectomy System — The device is indicated for mechanical de-clotting and controlled and selective infusion of physician specified fluids, including thrombolytics, in the peripheral vasculature.

SUMMARY:
This is an open label, prospective, non-randomised, multi-centre post market study of the POUNCE Venous Thrombectomy system for de-clotting in the peripheral vasculature (e.g., iliofemoral veins).

DETAILED DESCRIPTION:
This PMCF study is designed to further evaluate the safety and performance of the POUNCE Venous Thrombectomy system in the treatment of patients with symptomatic peripheral vascular thrombus through removal of thrombus. The study will collect both qualitative and quantitative data recorded by the investigators during the procedure to further evaluate safety and performance of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 years or older
2. Patients with peripheral vascular thrombus (e.g., iliofemoral) as confirmed by Doppler Ultrasonography (DUS)
3. Voluntary informed written consent, given before performance of any clinical investigation-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care
4. Patients who would likely experience benefit from mechanical thrombus removal

Exclusion Criteria:

1. Presence of a stent in the target vein
2. Known aggressive hypercoagulable states such as antiphospholipid antibody syndrome, Protein C/S Deficiency, Antithrombin deficiency, homozygous prothrombin gene mutation or homozygous Factor V Leiden
3. Limb-threatening circulatory compromise
4. Known symptomatic Pulmonary Embolism at the time of enrollment with or without severe RV dysfunction
5. Patients with a positive COVID test result at the time of the procedure
6. Patients who, according to the investigator, have a venous thrombus that may be associated with a prior COVID infection
7. History of, or active heparin induced thrombocytopenia (HIT)
8. Inability to withstand endovascular procedures
9. Life expectancy < 1 year
10. Participation in any other drug or device studies that have not reached the primary endpoint follow up, which could compromise the results of either trial
11. Patient has any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol
12. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel
13. Known or suspected abuse of alcohol, narcotics or non-prescription drugs that would jeopardize study outcomes in the Investigator's opinion
14. Inability to provide informed consent or to comply with study assessments (e.g., due to cognitive impairment or geographic distance)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Device Performance | 30 days, 1 year
  Successful preparation and use of the device to achieve flow restoration, i.e., elimination of a minimum of 50% thrombus (SIR Grade II or Grade III) in the treated target venous segment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, MD, Principal Investigator — Klinikum Hochsauerland GmbH

IPD SHARING:
Plan to Share IPD: Undecided